CLINICAL TRIAL: NCT00220597
Title: Group Interventions to Prevent HIV in High Risk Women
Brief Title: Group Therapies for Reducing HIV-risk Behavior in Women Who Have Survived Childhood Sexual Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Spiegel, Jack, Lulu & Sam Willson Professor, Stanford University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: R01MH060556 (NIH); R01MH060556 (NIH); DAHBR AZ-Q
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Alcoholism; Child Abuse, Sexual; Sexual Abuse; Sexual Behavior; Sexually Transmitted Diseases, Viral
Keywords: group therapy; sexual revictimization; risky sex; addiction
MeSH Terms: conditions — Alcoholism; Coitus; Sexual Behavior; Sexually Transmitted Diseases, Viral; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Trauma-focused group therapy

SUMMARY:
This study will evaluate the effectiveness of trauma-focused group therapy for reducing HIV-risk behavior and revictimization among adult women survivors of childhood sexual abuse (CSA).

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate the effectiveness of trauma-focused group therapy for reducing HIV risk behavior and revictimization among adult women survivors of childhood sexual abuse (CSA). Research indicates that childhood sexual abuse is a major risk factor for becoming HIV-infected. Individuals with CSA may be less able to benefit from HIV/AIDS prevention intervention if they are continuing to be traumatized by their earlier CSA experiences that interfere with their learning safer patterns of interpersonal and personal functioning. This study will examine whether or not it is helpful to focus on survivors' memories of CSA in order to reduce HIV risk behavior, revictimization, and distress. It will also examine potential mediators of treatment effectiveness for CSA survivors. This randomized clinical intervention trial will compare trauma-focused group therapy against a present-focused group therapy comparison condition and a case-management only control condition. All three groups will be provided with case management. We will recruit a total of 192 adult women survivors of childhood sexual abuse through newspaper advertisements and through local community organizations (e.g., community health clinics, rape crisis centers). All 192 research participants will meet criteria for posttraumatic stress disorder (PTSD) for CSA as well as have engaged in HIV risk behavior and/or experienced sexual revictimization within the past 3 months. These research participants will be recruited for a randomized clinical intervention trial to evaluate the effectiveness of the trauma-focused and present-focused treatment conditions and to identify mediators of treatment effects. Women for the randomized clinical intervention trial will be recruited in eight cohorts of 24 subjects each for randomization to treatment condition (trauma-focused or present-focused or case management only). Intervention subjects will be assessed on behavioral and other psychosocial measures at baseline and at 3-, 6-, 9-, and 12-month follow-up assessments to evaluate the effectiveness of trauma-focused treatment against the present-focused treatment and the case management only control condition in reducing HIV risk behavior, sexual revictimization, and trauma symptoms, and improving interpersonal functioning. We will examine three mediators of treatment effectiveness, including: 1) trauma reactive and resilient beliefs about self and the world; 2) differentiation and integration of self; and 3) interpersonal relations.

ELIGIBILITY:
Inclusion Criteria:

* 1. Female. 2. 18 years of age or older. 3. English-speaking. 4. Has at least two explicit memories of sexual abuse that involved genital contact.

  5. At least two sexual abuse events occurred when the survivor was between 4 and15 years of age.

  6. The perpetrator was at least 5 years older than the survivor. 7. The survivor knew the perpetrator prior to the sexual abuse. 8. The survivor has discussed or attempted to discuss details of the sexual abuse previously with another person (e.g., family member, friend, or therapist) at least 6 months prior to being interviewed for the study.

  9. Meets DSM-IV criteria for current PTSD. 10. Provides informed consent.

And at least one of the following:

11. Has been sexually revictimized within the previous year. 12. Has engaged in risky sexual behavior within the previous year. 13. Meets DSM-IV criteria for substance abuse

Exclusion Criteria:

* Criteria for exclusion includes any of the following:

  1. Diagnosed as meeting one of the following diagnostic categories: schizophrenia and other psychotic disorders; dementia and delirium and amnestic or other cognitive disorders.
  2. Reports ritual abuse.
  3. Is currently receiving psychotherapy (including individual or group psychotherapy).
  4. Individuals who are alcohol or drug dependent as defined by the DSM-IV.
  5. Individuals who are currently suicidal (i.e. within the last month)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 1999-09; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Rates of using of drugs or alcohol
Sexual revictimization rates
Rates of engaging in risky sex
Trauma symptoms

CONTACTS AND LOCATIONS:
Overall Officials: David Spiegel, M.D., Principal Investigator — Stanford University; Catherine C. Classen, Ph.D., Study Director — Stanford University
Locations (1):
- Dept. of Psychiatry, Stanford University, Stanford, California, United States